CLINICAL TRIAL: NCT06068959
Title: Effect of Photobiomodulation With LED Cluster on Pain and Mandibular and Cervical Mobility in Patients With Temporomandibular Dysfunction: Clinical, Randomized, Controlled and Blind Study
Brief Title: Photobiomodulation on Pain in Patients With Temporomandibular Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Anna Carolina Ratto Tempestini Horliana, Principal investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 220824a
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-09

CONDITIONS: TMJ Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation (Experimental): Photobiomodulation using a LED cluster
  Interventions: Device: Photobiomodulation using LED
- Placebo Photobiomodulation (Placebo Comparator): Placebo Photobiomodulation with the equipment turned off
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Photobiomodulation using LED — Photobiomodulation Using a Cluster of LEDs in the Red and Infrared Wavelengths in the Cervical Spine Region and Over the Masticatory Muscles
  Arms: Photobiomodulation
Device: Placebo — Photobiomodulation Placebo
  Arms: Placebo Photobiomodulation

SUMMARY:
These studies aim to validate the effects of photobiomodulation using clusters of 850nm LEDs (infrared) and 630nm LEDs (red); in pain and cervical and mandibular mobility in patients with TMD. It is a randomized, controlled, and blind clinical trial, which will consist of n= 36, of both genders, with ages ranging from 18 to 45 years, divided into 2 groups: Group 1 Red and infrared LED cluster, Group 2 placebo. The areas where they will receive photobiomodulation will be the TMJ area, masseter muscles, temporal muscles, scalenes, and trapezius. 6 non-consecutive sessions will be performed over 2 weeks. Diagnostic Criteria for Temporomandibular Disorders - DC/TMD will be used to determine TMD and validate participants. To validate the mandibular range of motion (ADM) a pachymeter will be used and for the cervical ADM a goniometer (fleximeter). The pain will be validated using the visual analog scale-VAS. All participants will be evaluated after the first therapeutic intervention, and again at the end, following the same validation procedures used initially.

DETAILED DESCRIPTION:
The term temporomandibular disorders (TMD), according to the American American Dental Association (ADA), refers to a group of disorders characterized by pain in the temporomandibular joint (TMD) in the periauricular area or in the masticatory muscles, in addition to TMD sounds during jaw function and deviation or restriction of jaw movements. Its multifactorial etiology is related to a heterogeneous group of functional, structural, and psychological factors, making it difficult to identify the association between a single etiological factor and the signs and symptoms of TMD. As a treatment option, it hasphotobiomodulation, using different light sources, alone or in combination. These studies aim to validate the effects of photobiomodulation using clusters of 850nm LEDs (infrared) and 630nm LEDs (red); in pain and cervical and mandibular mobility in patients with TMD. It is a randomized, controlled, and blind clinical trial, which will consist of n= 36, of both genders, with ages ranging from 18 to 45 years, divided into 2 groups: Group 1 Red and infrared LED cluster, Group 2 placebo. The areas where they will receive photobiomodulation will be the TMJ area, masseter muscles, temporal muscles, scalenes, and trapezius. 6 non-consecutive sessions will be performed over 2 weeks. Diagnostic Criteria for Temporomandibular Disorders - DC/TMD will be used to determine TMD and validate participants. To validate the mandibular range of motion (ADM) a pachymeter will be used and for the cervical ADM a goniometer (fleximeter). The pain will be validated using the visual analog scale-VAS. All participants will be evaluated after the first therapeutic intervention, and again at the end, following the same validation procedures used initially.

ELIGIBILITY:
Inclusion Criteria:

* present TMD according Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD) Axis I
* have all permanent teeth

Exclusion Criteria:

* be undergoing orthodontic treatment
* be undergoing other treatment for TMD
* present dental caries or gingival disease.
* Initiate or use any type of medication during the phases of the study
* comorbidity

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-02-29 (Estimated); Primary Completion 2024-07-10 (Estimated); Study Completion 2024-08-10 (Estimated)

PRIMARY OUTCOMES:
Pain Baseline | Before an intervention
  Evaluation of Pain using visual analogic scale in centimeters (0-10cm)
Final Pain | 2 weeks after treatment
  Evaluation of Pain using visual analogic scale in centimeters (0-10cm)

SECONDARY OUTCOMES:
Cervical spine mobility baseline | Before an intervention
  Evaluation of cervical spine mobility using goniometer in degrees
Final Cervical spine mobility | 2 weeks after intervention
  Evaluation of cervical spine mobility using goniometer in degrees
Mandibular mobility baseline | Before an intervention
  Evaluation of mandibular mobility using caliper in millimeters
Final Mandibular mobility | 2 weeks after intervention
  Evaluation of mandibular mobility using caliper in millimeters